CLINICAL TRIAL: NCT05029752
Title: Feasibility of Digital Thermal Monitoring to Assess Endothelium-Dependent Vasodilation in Patients Undergoing Hematopoietic Cell Transplantation (HCT)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: <75% participation
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-1309; NCI-2021-09419 (Other: NCI-CTRP Clinical Trials Process Registry)
Record Dates: First submitted 2021-08-25; First posted 2021-09-01 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Vascular; Endothelial; Endothelial Dysfunction; Endothelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Vendys II Device (Other): Your participation in this study will be over after your blood vessel health is measured 1 time with the Vendys II device
  Interventions: Device: Vendys II Device

INTERVENTIONS:
Device: Vendys II Device — Using the device

SUMMARY:
The Vendys II, an FDA-approved device, uses finger digital thermal monitoring (DTM) after a period of blood flow restriction to evaluate vascular health. This study will evaluate the feasibility of using this device to measure the Vascular Reactivity Index (VRI) in children and adolescents/young adults (AYA) undergoing hematopoietic cell transplantation (HCT).

DETAILED DESCRIPTION:
Primary Objective:

-Assess the feasibility of the use of VENDYS-II in children and AYA as a measure of vascular endothelial function, where feasibility is defined as completion of the evaluation by at least 70% of consented participants.

Secondary Objective:

-Summarize the incidence of any adverse events that precludes completion of assessment of endothelium-dependent vasodilation using the Vendys II in children and AYA.

ELIGIBILITY:
Inclusion Criteria for HCT candidates:

* Children, adolescents and young adults (AYA) 6-26 years of age who are HCT candidates
* Recipients within 30 days prior to or within 14 days after autologous and allogeneic HCT.

  -. Any preparative regimen.
* Willing and eligible to enroll on PA19-0756

Inclusion Criteria for Healthy Donors:

- Healthy HCT donors between the ages of 6-26 years of age.

Exclusion Criteria:

* Any subject who does not consent/assent to participation.

  -. Any subject with an injury or deformation to the index finger which prevents proper fit of the device.
* Any subject with skin toxicity or neuropathy which prevents comfortable use of the device.

Ages: 6 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
The use of VENDYS-II in children and AYA as a measure of vascular endothelial function. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Keri Schadler, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2024-04-11): https://cdn.clinicaltrials.gov/large-docs/52/NCT05029752/ICF_000.pdf